CLINICAL TRIAL: NCT00004730
Title: Magnesium Sulfate for Neuroprotection After Brain Trauma
Brief Title: Magnesium Sulfate For Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Nancy Temkin, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS019643 (NIH); NCT00004484 (obsolete NCT alias)
Record Dates: First submitted 2000-02-25; First posted 2000-02-28 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Brain Injuries; Head Injury; Brain Concussion
Keywords: head injury; traumatic brain injury; concussion; magnesium sulfate; neuroprotection
MeSH Terms: conditions — Brain Injuries; Craniocerebral Trauma; Brain Concussion; Brain Injuries, Traumatic | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: magnesium sulfate

SUMMARY:
The purpose of the study is to determine whether magnesium sulfate, given within 8 hours of a moderate or severe traumatic brain injury improves survival, decreases the number of people developing seizures, improves the survivors' mental and psychological functioning, including the ability to return to daily life, live independently, and return to work or school.

DETAILED DESCRIPTION:
The purpose of the study is to determine if treating head-injured patients with magnesium sulfate will improve medical, mental, and psychological recovery. In particular, the study will assess each patient's ability to return to daily life, live independently, and return to work or school as done before the head injury occurred. The study will also assess magnesium sulfate's ability to reduce the risk of developing seizures (epilepsy) as well as to improve survival rates after a traumatic brain injury. Patients on the study are assigned randomly (by chance) to either the magnesium sulfate group or the group which gets a placebo. This means they have an equal chance of being in either group. Before the first dose is given, two teaspoons worth of blood are drawn from a vein in the arm. The first dose of magnesium sulfate is 1meq/kg given intravenously within 8 hours of injury. Then a five day continuous intravenous infusion of magnesium sulfate 0.24meq/kg per hour is begun. Daily magnesium levels are checked and the dose changed in order to keep the Magnesium blood level at approximately 4meq/L. If the person does not receive magnesium sulfate, he receives a placebo which looks just like magnesium sulfate but contains no active medication. If the person leaves the hospital before the five days are over, the magnesium or placebo is stopped. Patients on the study will receive a brief exam in person or over the phone at one and three months after the injury to determine whether they have had any seizures and to evaluate how they are functioning and recovering from their head injury. Each evaluation will last about one hour. At six months after the injury, they will have full neuropsychological and psychosocial evaluations done at Harborview. These tests will take about five hours to complete and include tests of vocabulary, problem solving, and coordination. There will be questions about how the injury has affected the way they feel and interact socially. For example, there will be questions about their ability to work, manage personal affairs, what their moods are like, and how anger is handled.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury with post-resuscitation Glasgow Coma Scale of 3-12 or, if intubated, motor score of 1-5, or who require emergent neurosurgical intervention precluding the accurate assessment of Glasgow Coma Scale.

Exclusion Criteria:

* Injury greater than 8 hours old
* Age under 14 years
* Compromised renal function (creatinine of 2.0 mb/dl or greater)
* Membership in a vulnerable population (e.g. pregnant woman, prisoner, etc.)
* Residence making follow-up unlikely (e.g. lives outside U.S.)
* Refusal to participate

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Temkin, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Temkin NR, Anderson GD, Winn HR, Ellenbogen RG, Britz GW, Schuster J, Lucas T, Newell DW, Mansfield PN, Machamer JE, Barber J, Dikmen SS. Magnesium sulfate for neuroprotection after traumatic brain injury: a randomised controlled trial. Lancet Neurol. 2007 Jan;6(1):29-38. doi: 10.1016/S1474-4422(06)70630-5. PMID 17166799